CLINICAL TRIAL: NCT04833413
Title: Effectiveness of Regimen Switch After Intensive Insulin Therapy in Hospitalized Patients With Type 2 Diabetes
Brief Title: Regimen Switch After Intensive Insulin Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZSE-202104
Record Dates: First submitted 2021-04-03; First posted 2021-04-06 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Continue intensive treatment group: Patients with type 2 diabetes who continued intensive treatment within 6 months after hospital discharge
  Interventions: Drug: Continuous intensive insulin therapy
- Premixed insulin treatment group: Patients with type 2 diabetes who changed to premixed insulin within 6 months after hospital discharge
  Interventions: Drug: Continuous intensive insulin therapy
- Basic insulin treatment group: Patients with type 2 diabetes who changed to basic insulin treatment within 6 months after hospital discharge
  Interventions: Drug: Continuous intensive insulin therapy
- Oral hypoglycemic drug treatment group: Patients with type 2 diabetes who changed to oral hypoglycemic drug treatment within 6 months after hospital discharge

INTERVENTIONS:
Drug: Continuous intensive insulin therapy — After initial intensive insulin therapy in hospital, patients were grouped according to different treatment regimens within 6 months of discharge
  Other Names: Premixed insulin therapy; Basic insulin therapy; Oral hypoglycemic drug therapy
  Groups: Basic insulin treatment group; Continue intensive treatment group; Premixed insulin treatment group

SUMMARY:
Insulin intensive therapy have traditionally been considered a sequential therapy in type 2 diabetes last choice, a number of guidelines and consensus recommendations insulin intensive therapy can be as obvious hyperglycemia in patients with newly diagnosed T2DM part of a line, a subset of patients after insulin intensive treatment target often need to change to other treatments, especially for senile diabetes patients, due to its self management ability, simplify the insulin solution is more urgent. Current clinical guidelines do not provide specific clinical guidance, such as the timing and method of switch after initial insulin intensive therapy. The purpose of this study was to explore the timing, suitable population and conversion methods of insulin regimens after treatment.

DETAILED DESCRIPTION:
Selecting initial insulin intensive therapy during the period of hospitalization in patients with type 2 diabetes, collect the basic information and biochemical information collection, including gender, age, duration of diabetes, intensive glucose-lowering treatment plan before treatment, diabetes complications, merger disease, smoking, drinking, height, weight, blood pressure, fasting glucose, glycosylated hemoglobin and glycosylated serum protein, insulin, c-peptide, liver and kidney function, blood lipid, blood routine, hypoglycemia is happening almost 1 month. Follow-up was conducted in January, March and June. Endocrinologists decide whether to continue the original hypoglycemic regimen or adjust it according to the glycemic control goals, islet β-cell function, diabetes complications, complications, hypoglycemia and other combination drugs, as well as patients' treatment willingness and compliance. To compare the timing of conversion of treatment regimens, the proportion of conversion to each regimen and the situation of reaching the standard, and to further analyze and compare the characteristics of people who switched to different regimens, in order to establish the basis for the selection of adjustment regimens after insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes;
* Patients who started intensive insulin therapy during hospitalization
* Age ≥18 years old

Exclusion Criteria:

* Type 1 diabetes, special type diabetes
* Acute complications of diabetes (diabetic ketoacidosis, hyperglycemia and hyperosmolarity)
* Severe infection
* pregnancy or planned pregnancy
* Participating in other clinical studies or trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2021.4 -- 2022.6 Adult patients with type 2 diabetes admitted to the endocrinology department of a level-2 or higher hospital and initiated intensive insulin therapy during hospitalization
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 1，3，6 months
  HbA1c in different conversion regimens

SECONDARY OUTCOMES:
The average blood glucose | 1，3，6 months
  The average blood glucose in different conversion regimens
Fasting blood glucose | 1，3，6 months
  Fasting blood glucose in different conversion regimens
Postprandial blood glucose | 1，3，6 months
  Postprandial blood glucose in different conversion regimens
Incidence of hypoglycemia | 1，3，6 months
  Incidence of hypoglycemia in different conversion regimens
Impact on body weight | 1，3，6 months
  Impact on body weight in different conversion regimens

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhongshan hospital, Shanghai, Shanghai Municipality
  - Department of Endocrinoogy, Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided
Clinical study Report may be shared

REFERENCES:
- [Result] Home PD, Dain MP, Freemantle N, Kawamori R, Pfohl M, Brette S, Pilorget V, Scherbaum WA, Vespasiani G, Vincent M, Balkau B. Four-year evolution of insulin regimens, glycaemic control, hypoglycaemia and body weight after starting insulin therapy in type 2 diabetes across three continents. Diabetes Res Clin Pract. 2015 May;108(2):350-9. doi: 10.1016/j.diabres.2015.01.030. Epub 2015 Jan 23. PMID 25825361
- [Result] Jin SM, Kim JH, Min KW, Lee JH, Ahn KJ, Park JH, Jang HC, Park SW, Lee KW, Won KC, Kim YI, Chung CH, Park TS, Lee JH, Lee MK. Basal-prandial versus premixed insulin in patients with type 2 diabetes requiring insulin intensification after basal insulin optimization: A 24-week randomized non-inferiority trial. J Diabetes. 2016 May;8(3):405-13. doi: 10.1111/1753-0407.12312. Epub 2015 Jun 29. PMID 25952532
- [Result] Weng J. Short-term intensive insulin therapy could be the preferred option for new onset Type 2 diabetes mellitus patients with HbA1c > 9. J Diabetes. 2017 Oct;9(10):890-893. doi: 10.1111/1753-0407.12581. Epub 2017 Aug 22. PMID 28661564
- [Result] Davies MJ, D'Alessio DA, Fradkin J, Kernan WN, Mathieu C, Mingrone G, Rossing P, Tsapas A, Wexler DJ, Buse JB. Management of Hyperglycemia in Type 2 Diabetes, 2018. A Consensus Report by the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2018 Dec;41(12):2669-2701. doi: 10.2337/dci18-0033. Epub 2018 Oct 4. PMID 30291106
- [Result] Bellido V, Suarez L, Rodriguez MG, Sanchez C, Dieguez M, Riestra M, Casal F, Delgado E, Menendez E, Umpierrez GE. Comparison of Basal-Bolus and Premixed Insulin Regimens in Hospitalized Patients With Type 2 Diabetes. Diabetes Care. 2015 Dec;38(12):2211-6. doi: 10.2337/dc15-0160. Epub 2015 Oct 12. PMID 26459273
- [Result] Mauricio D, Meneghini L, Seufert J, Liao L, Wang H, Tong L, Cali A, Stella P, Carita P, Khunti K. Glycaemic control and hypoglycaemia burden in patients with type 2 diabetes initiating basal insulin in Europe and the USA. Diabetes Obes Metab. 2017 Aug;19(8):1155-1164. doi: 10.1111/dom.12927. Epub 2017 Apr 10. PMID 28251792
- [Result] Russell-Jones D, Pouwer F, Khunti K. Identification of barriers to insulin therapy and approaches to overcoming them. Diabetes Obes Metab. 2018 Mar;20(3):488-496. doi: 10.1111/dom.13132. Epub 2017 Nov 22. PMID 29053215
- [Result] Bowering K, Case C, Harvey J, Reeves M, Sampson M, Strzinek R, Bretler DM, Bang RB, Bode BW. Faster Aspart Versus Insulin Aspart as Part of a Basal-Bolus Regimen in Inadequately Controlled Type 2 Diabetes: The onset 2 Trial. Diabetes Care. 2017 Jul;40(7):951-957. doi: 10.2337/dc16-1770. Epub 2017 May 8. PMID 28483786
- [Result] Lind M, Hirsch IB, Tuomilehto J, Dahlqvist S, Ahren B, Torffvit O, Attvall S, Ekelund M, Filipsson K, Tengmark BO, Sjoberg S, Pehrsson NG. Liraglutide in people treated for type 2 diabetes with multiple daily insulin injections: randomised clinical trial (MDI Liraglutide trial). BMJ. 2015 Oct 28;351:h5364. doi: 10.1136/bmj.h5364. PMID 26512041
- [Result] American Diabetes Association. 15. Diabetes Care in the Hospital: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S211-S220. doi: 10.2337/dc21-S015. PMID 33298426